CLINICAL TRIAL: NCT02058147
Title: A Randomized, 30 Week, Active-controlled, Open-label, 3-treatment Arm, Parallel-group Multicenter Study Comparing the Efficacy and Safety of Insulin Glargine/ Lixisenatide Fixed Ratio Combination to Insulin Glargine Alone and to Lixisenatide Alone on Top of Metformin in Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Efficacy and Safety of Insulin Glargine/ Lixisenatide Fixed Ratio Combination Compared to Insulin Glargine Alone and Lixisenatide Alone on Top of Metformin in Patients With T2DM
Acronym: LixiLan-O
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12404; 2013-003131-30 (EudraCT Number); U1111-1148-4334 (Other: UTN)
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) (Experimental): FRC once daily (QD) for 30 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine/lixisenatide Fixed Ratio Combination; Drug: Metformin
- Insulin Glargine (Active Comparator): Insulin glargine QD for 30 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Metformin
- Lixisenatide (Active Comparator): Lixisenatide 10 mcg QD for 2 weeks, then 20 mcg QD (maintenance dose).
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Metformin

INTERVENTIONS:
Drug: Insulin glargine/lixisenatide Fixed Ratio Combination — Insulin glargine/Lixisenatide FRC was self-administered by subcutaneous (SC) injection in the morning within one hour before breakfast using one of the 2 prefilled disposable SoloStar® pen-injectors: Pen A containing 100 U/mL insulin glargine (Lantus, 100 U/mL) and 50 mcg/mL lixisenatide in a ratio of 2 U:1 mcg, used for administration of doses from 10 U to 40 U (10 U/5mcg to 40 U/20mcg). Pen B containing 100 U/mL insulin glargine (Lantus, 100 U/mL) and 33 mcg/mL lixisenatide in a ratio of 3 U:1 mcg, used to administer doses from 41 U to 60 U (41 U/13 mcg to 60 U/20 mcg). The starting dose was 10 U/5 mcg. Dose was then adjusted individually to reach and maintain fasting self-monitored plasma glucose (SMPG) of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L) while avoiding hypoglycemia.
  Other Names: (HOE901/AVE0010)
  Arms: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Drug: Insulin glargine (HOE901) — Insulin glargine (100 U/mL) was self-administered by SC injection at approximately the same time every day. Dose was adjusted individually to reach and maintain fasting SMPG of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L) while avoiding hypoglycemia.
  Other Names: Lantus
  Arms: Insulin Glargine
Drug: Lixisenatide (AVE0010) — Lixisenatide was self-administered by SC injection within 0 to 60 minutes before breakfast or evening meal. If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 10 mcg.
  Other Names: Lyxumia
  Arms: Lixisenatide
Drug: Metformin — Pharmaceutical form: Tablet; Route of administration: Oral administration.

SUMMARY:
Primary Objective:

To compare the insulin glargine/lixisenatide fixed ratio combination to lixisenatide alone and to insulin glargine alone (on top of metformin treatment) in glycated hemoglobin (HbA1c) change from baseline to Week 30.

Secondary Objective:

To compare the overall efficacy and safety of insulin glargine/lixisenatide fixed ratio combination (FRC) to insulin glargine alone and to lixisenatide alone (on top of metformin treatment) over a 30 week treatment period in participants with type 2 diabetes.

DETAILED DESCRIPTION:
Approximately 37 weeks including up to 6 weeks of screening, 30-week treatment period, and a 3 days follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Participants with type 2 diabetes mellitus diagnosed for at least 1 year before the screening visit, treated for at least 3 months prior to visit 1 with metformin alone or metformin and a second oral anti-diabetic treatment that could be a sulfonylurea, a glinide, a sodium glucose co-transporter-2 inhibitor or a di-peptidyl peptidase 4 (DPP-4) inhibitors, and who were not adequately controlled with this treatment.
* Signed written informed consent.

Exclusion criteria:

* HbA1c at screening visit:

  * less than 7.5% or more than 10% for participants previously treated with metformin alone,
  * less than 7.0% or more than 9% for participants previously treated with metformin and a second oral anti-diabetic treatment.
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Use of oral glucose-lowering agents other than those stated in the inclusion criteria or any injectable glucose-lowering agents during the 3 months before screening.
* Previous Treatment with insulin (except for short-term treatment due to intercurrent illness including gestational diabetes, at the discretion of the trial physician).
* History of discontinuation of a previous treatment with a glucagon-like peptide (GLP-1) receptor agonist (GLP-1 RA) due to safety/tolerability issue or lack of efficacy.
* Participant who previously participated in any clinical trial with lixisenatide or the insulin glargine/lixisenatide fixed ratio combination or had previously received lixisenatide.
* Any contraindication to metformin use, according to local labeling.
* Use of weight loss drugs within 3 months prior to screening visit.
* Within the last 6 months prior to screening visit: history of stroke, myocardial infarction, unstable angina, or heart failure requiring hospitalization. Planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy was already performed), chronic pancreatitis, pancreatitis during a previous treatment with incretin therapies, pancreatectomy, stomach/gastric surgery.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (e.g, multiple endocrine neoplasia syndromes).
* Uncontrolled or inadequately controlled hypertension (systolic blood pressure above 180 mmHg or diastolic blood pressure above 95 mmHg) at screening visit.
* At screening visit, Body Mass Index (BMI) less than or equal to 20 or above 40 kg/m^2.
* At screening visit amylase and/or lipase more than 3 times the upper limit of the normal (ULN) laboratory range.
* At screening visit alanine aminotransferase (ALT) or alkaline phosphatase (AST) more than 3 ULN.
* At screening visit calcitonin above or equal to 20 pg/mL (5.9 pmol/L).

Exclusion Criteria for randomization at the end of the screening period:

* HbA1c less than 7% or above 10%;
* Fasting Plasma glucose above 250 mg/dL (13.9 mmol/L);
* Metformin maximal tolerated dose less than 1500 mg/day;
* Amylase and/or lipase more than 3 ULN.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (273):
- United States (118):
  - Investigational Site Number 840027, Phoenix, Arizona
  - Investigational Site Number 840122, Phoenix, Arizona
  - Investigational Site Number 840062, Tempe, Arizona
  - Investigational Site Number 840023, Tempe, Arizona
  - Investigational Site Number 840084, Little Rock, Arkansas
  - Investigational Site Number 840100, Anaheim, California
  - Investigational Site Number 840065, Bell Gardens, California
  - Investigational Site Number 840090, Chino, California
  - Investigational Site Number 840002, Chula Vista, California
  - Investigational Site Number 840013, Concord, California
  - Investigational Site Number 840053, Fresno, California
  - Investigational Site Number 840017, La Jolla, California
  - Investigational Site Number 840070, Lancaster, California
  - Investigational Site Number 840121, Long Beach, California
  - Investigational Site Number 840126, Los Angeles, California
  - Investigational Site Number 840044, Los Angeles, California
  - Investigational Site Number 840101, Mission Hills, California
  - Investigational Site Number 840086, Mission Viejo, California
  - Investigational Site Number 840120, Mission Viejo, California
  - Investigational Site Number 840005, Northridge, California
  - Investigational Site Number 840034, Palm Springs, California
  - Investigational Site Number 840074, Port Hueneme, California
  - Investigational Site Number 840068, San Ramon, California
  - Investigational Site Number 840067, Santa Ana, California
  - Investigational Site Number 840029, Tarzana, California
  - Investigational Site Number 840006, Temecula, California
  - Investigational Site Number 840078, West Hills, California
  - Investigational Site Number 840059, Aurora, Colorado
  - Investigational Site Number 840038, Denver, Colorado
  - Investigational Site Number 840104, Bradenton, Florida
  - Investigational Site Number 840098, Miami, Florida
  - Investigational Site Number 840014, New Port Richey, Florida
  - Investigational Site Number 840047, Ocoee, Florida
  - Investigational Site Number 840056, Palm Harbor, Florida
  - Investigational Site Number 840089, Atlanta, Georgia
  - Investigational Site Number 840054, Lawrenceville, Georgia
  - Investigational Site Number 840119, Woodstock, Georgia
  - Investigational Site Number 840108, Idaho Falls, Idaho
  - Investigational Site Number 840075, Arlington Heights, Illinois
  - Investigational Site Number 840080, Chicago, Illinois
  - Investigational Site Number 840026, Chicago, Illinois
  - Investigational Site Number 840116, Chicago, Illinois
  - Investigational Site Number 840050, Springfield, Illinois
  - Investigational Site Number 840008, Avon, Indiana
  - Investigational Site Number 840015, Avon, Indiana
  - Investigational Site Number 840076, Avon, Indiana
  - Investigational Site Number 840082, Evansville, Indiana
  - Investigational Site Number 840031, Evansville, Indiana
  - Investigational Site Number 840060, Evansville, Indiana
  - Investigational Site Number 840048, Indianapolis, Indiana
  - Investigational Site Number 840085, Indianapolis, Indiana
  - Investigational Site Number 840012, Valparaiso, Indiana
  - Investigational Site Number 840025, Waterloo, Iowa
  - Investigational Site Number 840022, Lexington, Kentucky
  - Investigational Site Number 840007, Louisville, Kentucky
  - Investigational Site Number 840081, New Orleans, Louisiana
  - Investigational Site Number 840097, Auburn, Maine
  - Investigational Site Number 840063, Rockville, Maryland
  - Investigational Site Number 840028, Bloomfield Hills, Michigan
  - Investigational Site Number 840071, Chesterfield, Michigan
  - Investigational Site Number 840001, Dearborn, Michigan
  - Investigational Site Number 840091, Kalamazoo, Michigan
  - Investigational Site Number 840009, Minneapolis, Minnesota
  - Investigational Site Number 840024, Chesterfield, Missouri
  - Investigational Site Number 840057, Butte, Montana
  - Investigational Site Number 840042, Omaha, Nebraska
  - Investigational Site Number 840109, Henderson, Nevada
  - Investigational Site Number 840052, Las Vegas, Nevada
  - Investigational Site Number 840069, Nashua, New Hampshire
  - Investigational Site Number 840123, Morganville, New Jersey
  - Investigational Site Number 840011, Albuquerque, New Mexico
  - Investigational Site Number 840030, New Hyde Park, New York
  - Investigational Site Number 840096, Syracuse, New York
  - Investigational Site Number 840039, Asheville, North Carolina
  - Investigational Site Number 840021, Hickory, North Carolina
  - Investigational Site Number 840046, Morehead City, North Carolina
  - Investigational Site Number 840072, Morganton, North Carolina
  - Investigational Site Number 840110, Salisbury, North Carolina
  - Investigational Site Number 840095, Wilmington, North Carolina
  - Investigational Site Number 840099, Winston-Salem, North Carolina
  - Investigational Site Number 840004, Columbus, Ohio
  - Investigational Site Number 840016, Maumee, Ohio
  - Investigational Site Number 840103, Eugene, Oregon
  - Investigational Site Number 840113, Portland, Oregon
  - Investigational Site Number 840036, Pittsburgh, Pennsylvania
  - Investigational Site Number 840043, Tipton, Pennsylvania
  - Investigational Site Number 840058, Anderson, South Carolina
  - Investigational Site Number 840127, Charleston, South Carolina
  - Investigational Site Number 840049, Greer, South Carolina
  - Investigational Site Number 840114, Rapid City, South Dakota
  - Investigational Site Number 840112, Bristol, Tennessee
  - Investigational Site Number 840094, Knoxville, Tennessee
  - Investigational Site Number 840051, Austin, Texas
  - Investigational Site Number 840066, Corpus Christi, Texas
  - Investigational Site Number 840111, Dallas, Texas
  - Investigational Site Number 840020, Dallas, Texas
  - Investigational Site Number 840064, Dallas, Texas
  - Investigational Site Number 840003, Dallas, Texas
  - Investigational Site Number 840088, Edinburg, Texas
  - Investigational Site Number 840118, Fort Worth, Texas
  - Investigational Site Number 840055, Houston, Texas
  - Investigational Site Number 840087, Houston, Texas
  - Investigational Site Number 840079, Hurst, Texas
  - Investigational Site Number 840073, N Richland Hill, Texas
  - Investigational Site Number 840019, San Antonio, Texas
  - Investigational Site Number 840037, Draper, Utah
  - Investigational Site Number 840093, Ogden, Utah
  - Investigational Site Number 840061, Salt Lake City, Utah
  - Investigational Site Number 840041, Salt Lake City, Utah
  - Investigational Site Number 840040, Chesapeake, Virginia
  - Investigational Site Number 840045, Norfolk, Virginia
  - Investigational Site Number 840092, Norfolk, Virginia
  - Investigational Site Number 840125, Richmond, Virginia
  - Investigational Site Number 840115, Salem, Virginia
  - Investigational Site Number 840010, Weber City, Virginia
  - Investigational Site Number 840077, Federal Way, Washington
  - Investigational Site Number 840102, Renton, Washington
  - Investigational Site Number 840033, Milwaukee, Wisconsin
- Australia (4):
  - Investigational Site Number 036005, Box Hill
  - Investigational Site Number 036001, Camperdown
  - Investigational Site Number 036006, Kippa-Ring
  - Investigational Site Number 036007, Logan Central
- Belgium (3):
  - Investigational Site Number 056005, Brussels
  - Investigational Site Number 056006, Brussels
  - Investigational Site Number 056001, Leuven
- Canada (3):
  - Investigational Site Number 124004, Kelowna
  - Investigational Site Number 124001, Toronto
  - Investigational Site Number 124002, Vancouver
- Chile (11):
  - Investigational Site Number 152008, Osorno
  - Investigational Site Number 152015, Puerto Varas
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152006, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152012, Santiago
  - Investigational Site Number 152009, Santiago
  - Investigational Site Number 152011, Talagante
  - Investigational Site Number 152014, Temuco
  - Investigational Site Number 152003, Temuco
- Czechia (13):
  - Investigational Site Number 203004, Beroun
  - Investigational Site Number 203008, České Budějovice
  - Investigational Site Number 203014, Hořovice
  - Investigational Site Number 203012, Kopřivnice
  - Investigational Site Number 203001, Pardubice
  - Investigational Site Number 203005, Pilsen
  - Investigational Site Number 203003, Prague
  - Investigational Site Number 203009, Prague
  - Investigational Site Number 203007, Prague
  - Investigational Site Number 203013, Praha 9 - Klanovice
  - Investigational Site Number 203006, Trutnov
  - Investigational Site Number 203016, Újezd u Brna
  - Investigational Site Number 203015, Vsetín
- Denmark (6):
  - Investigational Site Number 208003, Aarhus C
  - Investigational Site Number 208009, Horsens
  - Investigational Site Number 208002, Kolding
  - Investigational Site Number 208001, København NV
  - Investigational Site Number 208005, København S
  - Investigational Site Number 208004, Viborg
- Estonia (4):
  - Investigational Site Number 233004, Paide
  - Investigational Site Number 233002, Pärnu
  - Investigational Site Number 233003, Tallinn
  - Investigational Site Number 233001, Viljandimaa
- France (4):
  - Investigational Site Number 250006, Corbeil-Essonnes
  - Investigational Site Number 250002, La Rochelle
  - Investigational Site Number 250003, Pierre-Bénite
  - Investigational Site Number 250001, Vénissieux
- Germany (7):
  - Investigational Site Number 276005, Berlin
  - Investigational Site Number 276003, Berlin
  - Investigational Site Number 276004, Dortmund
  - Investigational Site Number 276007, Dresden
  - Investigational Site Number 276001, Dresden
  - Investigational Site Number 276006, Hamburg
  - Investigational Site Number 276002, Neumünster
- Hungary (10):
  - Investigational Site Number 348003, Balatonfüred
  - Investigational Site Number 348007, Budapest
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348011, Komárom
  - Investigational Site Number 348008, Nagykanizsa
  - Investigational Site Number 348012, Sátoraljaújhely
  - Investigational Site Number 348004, Szeged
  - Investigational Site Number 348010, Székesfehérvár
  - Investigational Site Number 348001, Zalaegerszeg
- Italy (5):
  - Investigational Site Number 380002, Bologna
  - Investigational Site Number 380006, Catanzaro
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380003, Napoli
  - Investigational Site Number 380005, Roma
- Latvia (4):
  - Investigational Site Number 428002, Riga
  - Investigational Site Number 428003, Riga
  - Investigational Site Number 428004, Riga
  - Investigational Site Number 428001, Sigulda
- Lithuania (7):
  - Investigational Site Number 440003, Jonava
  - Investigational Site Number 440002, Kaunas
  - Investigational Site Number 440007, Kaunas
  - Investigational Site Number 440004, Kėdainiai
  - Investigational Site Number 440006, Panevezys
  - Investigational Site Number 440005, Utena
  - Investigational Site Number 440001, Vilnius
- Mexico (8):
  - Investigational Site Number 484005, Aguascalientes
  - Investigational Site Number 484001, Cuernavaca
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484004, Guadalajara
  - Investigational Site Number 484009, Guadalajara
  - Investigational Site Number 484007, Monterrey
  - Investigational Site Number 484006, Monterrey
  - Investigational Site Number 484010, Zapopan
- Poland (8):
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616005, Krakow
  - Investigational Site Number 616006, Krakow
  - Investigational Site Number 616007, Lodz
  - Investigational Site Number 616004, Szczecin
  - Investigational Site Number 616003, Warsaw
  - Investigational Site Number 616001, Warsaw
  - Investigational Site Number 616008, Żory
- Romania (9):
  - Investigational Site Number 642008, Bucharest
  - Investigational Site Number 642007, Bucharest
  - Investigational Site Number 642009, Cluj-Napoca
  - Investigational Site Number 642006, Hunedoara
  - Investigational Site Number 642005, Iași
  - Investigational Site Number 642002, Oradea
  - Investigational Site Number 642001, Târgu Mureş
  - Investigational Site Number 642004, Timișoara
  - Investigational Site Number 642003, Timișoara
- Russia (13):
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643008, Penza
  - Investigational Site Number 643012, Petrozavodsk
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643007, Saint Petersburg
  - Investigational Site Number 643003, Saint Petersburg
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643014, Samara
  - Investigational Site Number 643009, Saratov
  - Investigational Site Number 643011, Saratov
  - Investigational Site Number 643016, Tomsk
  - Investigational Site Number 643004, Voronezh
- South Africa (7):
  - Investigational Site Number 710002, Cap Town
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710005, Meyerspark
  - Investigational Site Number 710007, Port Elizabeth
  - Investigational Site Number 710004, Pretoria
  - Investigational Site Number 710001, Somerset West
  - Investigational Site Number 710006, Soweto
- Spain (11):
  - Investigational Site Number 724011, A Coruña
  - Investigational Site Number 724012, Barcelona
  - Investigational Site Number 724009, Granada
  - Investigational Site Number 724004, Hostalets de Balenyà
  - Investigational Site Number 724007, Lugo
  - Investigational Site Number 724008, Madrid
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724013, Palma de Mallorca
  - Investigational Site Number 724001, Quart de Poblet
  - Investigational Site Number 724006, Sant Joan Despí
  - Investigational Site Number 724003, Seville
- Sweden (5):
  - Investigational Site Number 752001, Ljungby
  - Investigational Site Number 752003, Malmo
  - Investigational Site Number 752004, Rättvik
  - Investigational Site Number 752005, Stockholm
  - Investigational Site Number 752002, Vällingby
- Ukraine (8):
  - Investigational Site Number 804002, Chernivtsi
  - Investigational Site Number 804009, Ivano-Frankivsk
  - Investigational Site Number 804010, Kyiv
  - Investigational Site Number 804007, Kyiv
  - Investigational Site Number 804006, Kyiv
  - Investigational Site Number 804012, Lviv
  - Investigational Site Number 804011, Vinnytsia
  - Investigational Site Number 804008, Vinnytsia
- United Kingdom (5):
  - Investigational Site Number 826001, Coventry
  - Investigational Site Number 826002, Dundee
  - Investigational Site Number 826006, Guildford
  - Investigational Site Number 826007, Leicester
  - Investigational Site Number 826003, Norwich

REFERENCES:
- [Result] Rosenstock J, Aronson R, Grunberger G, Hanefeld M, Piatti P, Serusclat P, Cheng X, Zhou T, Niemoeller E, Souhami E, Davies M; LixiLan-O Trial Investigators. Benefits of LixiLan, a Titratable Fixed-Ratio Combination of Insulin Glargine Plus Lixisenatide, Versus Insulin Glargine and Lixisenatide Monocomponents in Type 2 Diabetes Inadequately Controlled on Oral Agents: The LixiLan-O Randomized Trial. Diabetes Care. 2016 Nov;39(11):2026-2035. doi: 10.2337/dc16-0917. Epub 2016 Aug 15. PMID 27527848
- [Derived] Shao H, Kianmehr H, Guo J, Li P, Fonseca V, Shi L. Efficacy of iGlarLixi on 5-year risk of diabetes-related complications: A simulation study. J Diabetes Complications. 2022 Mar;36(3):108132. doi: 10.1016/j.jdiacomp.2022.108132. Epub 2022 Jan 25. PMID 35101326
- [Derived] Davies MJ, Russell-Jones D, Barber TM, Lavalle-Gonzalez FJ, Galstyan GR, Zhu D, Baxter M, Dessapt-Baradez C, McCrimmon RJ. Glycaemic benefit of iGlarLixi in insulin-naive type 2 diabetes patients with high HbA1c or those with inadequate glycaemic control on two oral antihyperglycaemic drugs in the LixiLan-O randomized trial. Diabetes Obes Metab. 2019 Aug;21(8):1967-1972. doi: 10.1111/dom.13791. Epub 2019 Jun 18. PMID 31124299
- [Derived] Dailey G, Bajaj HS, Dex T, Groleau M, Stager W, Vinik A. Post hoc efficacy and safety analysis of insulin glargine/lixisenatide fixed- ratio combination in North American patients compared with the rest of world. BMJ Open Diabetes Res Care. 2019 Mar 21;7(1):e000581. doi: 10.1136/bmjdrc-2018-000581. eCollection 2019. PMID 31114694
- [Derived] Schmider W, Belder R, Lee M, Niemoeller E, Souhami E, Frias JP. Impact of dose capping in insulin glargine/lixisenatide fixed-ratio combination trials in patients with type 2 diabetes. Curr Med Res Opin. 2019 Jun;35(6):1081-1089. doi: 10.1080/03007995.2018.1558852. Epub 2019 Jan 11. PMID 30550345
- [Derived] Rosenstock J, Handelsman Y, Vidal J, Ampudia Blasco FJ, Giorgino F, Liu M, Perfetti R, Meier JJ. Propensity-score-matched comparative analyses of simultaneously administered fixed-ratio insulin glargine 100 U and lixisenatide (iGlarLixi) vs sequential administration of insulin glargine and lixisenatide in uncontrolled type 2 diabetes. Diabetes Obes Metab. 2018 Dec;20(12):2821-2829. doi: 10.1111/dom.13462. Epub 2018 Aug 13. PMID 29974618
- [Derived] Trujillo JM, Roberts M, Dex T, Chao J, White J, LaSalle J. Low incidence of gastrointestinal adverse events over time with a fixed-ratio combination of insulin glargine and lixisenatide versus lixisenatide alone. Diabetes Obes Metab. 2018 Nov;20(11):2690-2694. doi: 10.1111/dom.13444. Epub 2018 Aug 21. PMID 29923298
- [Derived] Davies MJ, Leiter LA, Guerci B, Grunberger G, Ampudia-Blasco FJ, Yu C, Stager W, Niemoeller E, Souhami E, Rosenstock J. Impact of baseline glycated haemoglobin, diabetes duration and body mass index on clinical outcomes in the LixiLan-O trial testing a titratable fixed-ratio combination of insulin glargine/lixisenatide (iGlarLixi) vs insulin glargine and lixisenatide monocomponents. Diabetes Obes Metab. 2017 Dec;19(12):1798-1804. doi: 10.1111/dom.12980. Epub 2017 Jul 7. PMID 28432746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 240 centers in 23 countries. A total of 2457 participants were screened between February 12, 2014 and September 16, 2014. 978 participants were not eligible for run-in mainly due to glycosylated hemoglobin (HbA1c) value at screening visit being out of the protocol defined range.
Pre-assignment Details: After 2 weeks screening period, 1479 participants underwent 4-week run-in period. 309 participants were run-in failures. A total of 1170 participants were randomized in 2:2:1 to insulin glargine/lixisenatide, insulin glargine and lixisenatide arms respectively in open-label treatment period.
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): FRC injected subcutaneously once daily (QD) for 30 weeks. Dose individually adjusted.
- Insulin Glargine: Insulin glargine injected subcutaneously QD for 30 weeks. Dose individually adjusted.
- Lixisenatide: Lixisenatide 10 mcg injected subcutaneously QD for 2 weeks, then 20 mcg QD (maintenance dose).
Period: Overall Study
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | Insulin Glargine | Lixisenatide
Started | 469 | 467 | 234
Treated | 469 | 467 | 233
Completed | 440 | 440 | 205
Not Completed | 29 | 27 | 29
Not completed — Randomized but not treated | 0 | 0 | 1
Not completed — Adverse Event | 12 | 9 | 21
Not completed — Lack of Efficacy | 1 | 0 | 3
Not completed — Poor compliance to protocol | 8 | 9 | 4
Not completed — Other than specified | 8 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 30 weeks. Dose individually adjusted.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide | Total
Number analyzed (Participants) | 469 | 467 | 234 | 1170
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.5) | 58.3 (9.4) | 58.7 (8.7) | 58.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 230 | 101 | 578
  Male | 222 | 237 | 133 | 592
Race [Count of Participants; unit: Participants]
  Caucasian | 417 | 421 | 216 | 1054
  Black | 33 | 33 | 12 | 78
  Asian/Oriental | 8 | 7 | 3 | 18
  Other | 11 | 6 | 3 | 20
Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 85 | 87 | 51 | 223
  Not Hispanic | 384 | 380 | 183 | 947
Second Oral Anti-diabetic Drug (OAD) Use [Count of Participants; unit: Participants]
  Yes | 274 | 270 | 133 | 677
  No | 195 | 197 | 101 | 493
Second OAD Use at Screening by Class [Count of Participants; unit: Participants]
  Sulfonylurea | 259 | 249 | 123 | 631
  Glinide | 3 | 10 | 5 | 18
  Sodium-glucose co-transporter-2 inhibitor | 2 | 2 | 0 | 4
  Dipeptidyl peptidase-4 inhibitor | 12 | 11 | 5 | 28
  None | 193 | 195 | 101 | 489
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.64 (4.4) | 31.66 (4.51) | 31.99 (4.39) | 31.72 (4.44)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.89 (5.51) | 8.66 (5.59) | 8.89 (6.26) | 8.80 (5.69)
Daily Dose of Metformin [Mean (Standard Deviation); unit: mg] | 2246.1 (456.8) | 2244.7 (444.7) | 2267.3 (427.4) | 2249.8 (445.9)
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.08 (0.71) | 8.08 (0.69) | 8.13 (0.72) | 8.09 (0.70)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.87 (2.35) | 9.75 (2.32) | 9.75 (2.19) | 9.80 (2.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 30
Description: Primary outcome was to test superiority of FRC versus Lixisenatide and non-inferiority versus Insulin glargine.
  Change in HbA1c was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: Modified intent-to-treat (mITT) population: all randomized participants who had both baseline and at least one post-baseline efficacy assessment. Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 467 | 464 | 233
percentage of hemoglobin | -1.63 (0.038) | -1.34 (0.039) | -0.85 (0.052)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Lixisenatide; Analysis was performed using Mixed-effect model with repeated measures (MMRM) with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline HbA1c value-by-visit interaction as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤0.05; Least Square (LS) Mean Difference = -0.78, 95% CI 2-sided [-0.898 to -0.665], Standard Error of Mean 0.059 — Insulin Glargine/Lixisenatide FRC vs Lixisenatide
Statistical Analysis 2: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline HbA1c value-by-visit interaction as a covariate; Test type: Non-Inferiority or Equivalence — Predefined non-inferiority margin of 0.3%; Mixed Models Analysis; LS Mean Difference = -0.29, 95% CI 2-sided [-0.384 to -0.194], Standard Error of Mean 0.048 — Insulin Glargine/Lixisenatide FRC vs Insulin glargine
Statistical Analysis 3: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Test of superiority was also performed as a secondary endpoint according to hierarchical testing procedure. Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline HbA1c value-by-visit interaction, as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -0.29, 95% CI 2-sided [-0.384 to -0.194], Standard Error of Mean 0.048 — Insulin Glargine/Lixisenatide FRC vs Insulin glargine

2. Secondary Outcome: Percentage of Participants With HbA1c <7.0% or ≤6.5% at Week 30
Description: Participants without Week 30 value for HbA1c were counted as non-responders.
Time Frame: Week 30
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 468 | 466 | 233
percentage of participants
  HbA1c <7.0% | 73.7 | 59.4 | 33
  HbA1c ≤6.5% | 55.8 | 39.5 | 19.3
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Lixisenatide; HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Lixisenatide. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of second OAD use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤0.05; Difference in percentage = 40.61, 95% CI 2-sided [33.63 to 47.59] — HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Lixisenatide
Statistical Analysis 2: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Lixisenatide; HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Lixisenatide. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of second OAD use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤ 0.05; Difference in percentage = 36.38, 95% CI 2-sided [29.81 to 42.95] — HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Lixisenatide
Statistical Analysis 3: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Insulin glargine. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of second OAD use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤ 0.05; Difference in percentage = 14.31, 95% CI 2-sided [8.37 to 20.25] — HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Insulin glargine
Statistical Analysis 4: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Insulin glargine. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of second OAD use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤ 0.05; Difference in percentage = 16.35, 95% CI 2-sided [10.13 to 22.58] — HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Insulin glargine

3. Secondary Outcome: Change in Plasma Glucose Excursion From Baseline to Week 30
Description: Plasma glucose excursion = 2-hour postprandial plasma glucose (PPG) value minus plasma glucose value obtained 30 minutes prior to the start of meal and before investigational medicinal product (IMP) administration if IMP was injected before breakfast. Change in plasma glucose excursions were calculated by subtracting baseline value from Week 30 value. Missing data was imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline plasma glucose excursion assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 428 | 425 | 192
mmol/L | -2.31 (0.154) | -0.18 (0.157) | -3.23 (0.216)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of Week -1 HbA1c (<8.0,≥8.0%), randomization strata of second OAD use at screening & country as fixed effects & baseline plasma glucose excursion value as a covariate. Hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially per pre-specified order; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤0.05. The hierarchical testing continued only when primary hypotheses (superiority: FRC to lixisenatide; non-inferiority: FRC to insulin glargine for HbA1c) was statistically significant; LS Mean Difference = -2.13, 95% CI 2-sided [-2.498 to -1.77], Standard Error of Mean 0.185 — Insulin Glargine/Lixisenatide FRC vs Insulin glargine

4. Secondary Outcome: Change in Body Weight From Baseline to Week 30
Description: Change in body weight was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline body weight assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 467 | 465 | 233
kg | -0.29 (0.182) | 1.11 (0.183) | -2.3 (0.256)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline body weight value-by-visit interaction as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -1.4, 95% CI 2-sided [-1.891 to -0.91], Standard Error of Mean 0.25 — Insulin Glargine/Lixisenatide FRC vs Insulin glargine

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 30
Description: Change in FPG was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analysed = participants with baseline and at least one post-baseline FPG assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 465 | 465 | 232
mmol/L | -3.46 (0.09) | -3.27 (0.091) | -1.5 (0.124)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Lixisenatide; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline FPG value-by-visit interaction as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -1.96, 95% CI 2-sided [-2.246 to -1.682], Standard Error of Mean 0.144 — Insulin Glargine/Lixisenatide FRC vs Lixisenatide

6. Secondary Outcome: Mean Change in 7-point Self-monitored Plasma Glucose (SMPG) Profile From Baseline to Week 30
Description: Participants recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime two times in a week before baseline, before visit Week 12 and before visit Week 30 and the average value across the profiles performed in the week before a visit for the 7-time points was calculated. Change in average 7-point SMPG was calculated by subtracting baseline value from Week 30 value. The analysis included all scheduled measurements obtained during the study. The missing data was handled by mixed effect model with repeated measures (MMRM) approach.
Time Frame: Baseline, Week 30
Population: mITT population. Here,number of participants analyzed = participants with baseline and at least one post baseline 7-point SMPG assessment during study period.
Measure: Least Squares Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 421 | 411 | 204
mmol/L | -3.35 (0.081) | -2.66 (0.084) | -1.95 (0.111)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Lixisenatide; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline 7-point SMPG value-by-visit interaction as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -1.4, 95% CI 2-sided [-1.645 to -1.158], Standard Error of Mean 0.124 — Insulin Glargine/Lixisenatide FRC vs Lixisenatide
Statistical Analysis 2: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects and baseline 7-point SMPG value-by-visit interaction, as a covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -0.69, 95% CI 2-sided [-0.892 to -0.495], Standard Error of Mean 0.101 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

7. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% With No Body Weight Gain at Week 30
Time Frame: Week 30
Population: mITT population. Participants without any HbA1c and/or body weight value at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 468 | 466 | 233
percentage of participants | 43.2 | 25.1 | 27.9
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8%, ≥8%) and randomization strata of second OAD use at screening; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤ 0.05; Difference in percentage = 18.08, 95% CI 2-sided [12.15 to 24.01] — Insulin Glargine/Lixisenatide FRC vs Insulin glargine

8. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% With No Body Weight Gain at Week 30 and No Documented Symptomatic Hypoglycemia (Plasma Glucose [PG] ≤ 70 mg/dL [3.9 mmol/L]) During 30-Week Treatment Period
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤70 mg/dL (3.9 mmol/L).
Time Frame: Baseline up to Week 30
Population: mITT population. Participants without any HbA1c and/or body weight value at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 468 | 466 | 233
percentage of participants | 31.8 | 18.9 | 26.2
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of second OAD use at screening; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance ≤ 0.05; Difference in percentage = 12.98, 95% CI 2-sided [7.5 to 18.45] — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

9. Secondary Outcome: Average Daily Insulin Glargine Dose at Week 30
Description: The analysis included scheduled measurements obtained up to the date of last injection of the IMP, including those obtained after introduction of rescue therapy.
Time Frame: Week 30
Population: mITT population. Here, number of participants analyzed = participants with insulin glargine dose assessment during study period. Data of this endpoint was planned to be analyzed for Insulin Glargine/Lixisenatide FRC and Insulin glargine arms only, not for lixisenatide arm.
Measure: Least Squares Mean (Standard Error); unit: Units (U)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 467 | 463
Units (U) | 39.77 (0.699) | 40.46 (0.701)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of second OAD use at screening, visits, treatment-by-visit interaction, and country as fixed effects; Test type: Superiority or Other; p = 0.4857, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -0.69, 95% CI 2-sided [-2.632 to 1.252], Standard Error of Mean 0.99 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

10. Secondary Outcome: Change in 2-Hour Postprandial Plasma Glucose (PPG) From Baseline to Week 30
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a liquid standardized breakfast meal. Change in PPG was calculated by subtracting baseline value from Week 30 value. Missing data was imputed using LOCF.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline 2-hour PPG assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 430 | 430 | 196
mmol/L | -5.68 (0.176) | -3.31 (0.178) | -4.58 (0.245)

11. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% at Week 30 With No Documented Symptomatic Hypoglycemia (PG ≤ 70 mg/dL [3.9 mmol/L]) During 30-Week Treatment Period
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤70 mg/dL (3.9 mmol/L). The analysis included all HbA1c measurements at Week 30, including those obtained after the IMP discontinuation or the introduction of rescue medication.
Time Frame: Baseline up to Week 30
Population: mITT population. Participants without Week 30 value for HbA1c were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 468 | 466 | 233
percentage of participants | 53.6 | 44.4 | 30.5

12. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During 30-Week Treatment Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after Week 12) was performed. Threshold values - from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 30: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8%.
Time Frame: Baseline up to Week 30
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 468 | 466 | 233
percentage of participants | 3.6 | 3.4 | 12.4

13. Secondary Outcome: Number of Documented Symptomatic Hypoglycemia Events Per Subject-Year
Description: Documented symptomatic hypoglycemia was an event during which symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤ 70 mg/dL (3.9 mmol/L).
Time Frame: First dose of study drug up to 1 day after the last dose administration (median treatment exposure: 211 days)
Population: Analysis was performed on safety population defined as all randomized participants who received at least one dose of IMP regardless of the amount of treatment administered.
Measure: Number; unit: Events per subject-year
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 469 | 467 | 233
Events per subject-year | 1.44 | 1.22 | 0.34

14. Secondary Outcome: Percentage of Participants With Documented Symptomatic Hypoglycemia
Description: as for outcome 13
Time Frame: First dose of study drug up to 1 day after the last dose administration (median treatment exposure: 211 days)
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 469 | 467 | 233
percentage of participants | 25.6 | 23.6 | 6.4

15. Secondary Outcome: Percentage of Participants With Severe Symptomatic Hypoglycemia
Description: Severe symptomatic hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Plasma glucose measurements might not have been available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal was considered sufficient evidence that the event had been induced by a low plasma glucose concentration. Severe symptomatic hypoglycemia included all episodes in which neurological impairment was severe enough to prevent self-treatment, and which were thus thought to place participants at risk of injury to themselves or others.
Time Frame: First dose of study drug up to 1 day after the last dose administration (median treatment exposure: 211 days)
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Number analyzed (Participants) | 469 | 467 | 233
percentage of participants | 0 | 0.2 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Day 213) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent that is AEs that developed/worsened during 'on-treatment period' (time from first injection of open-label IMP up to 3 days after the last injection of IMP regardless of the introduction of rescue therapy). Analysis was done on safety population.
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 30 weeks. Dose individually adjusted (median exposure: 211 days).
- Insulin Glargine: Insulin glargine injected subcutaneously QD for 30 weeks. Dose individually adjusted (median exposure: 211 days).
- Lixisenatide: Lixisenatide 10 mcg injected subcutaneously QD for 2 weeks, then 20 mcg QD (maintenance dose) median exposure: 211 days).
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 18/469 | 19/467 | 9/233
Other Adverse Events (participants affected / at risk) | 138/469 | 85/467 | 98/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=469) | Insulin Glargine (N=467) | Lixisenatide (N=233)
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Meningitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=469) | Insulin Glargine (N=467) | Lixisenatide (N=233)
Upper respiratory tract infection (Infections and infestations) | 33 | 23 | 12
Nasopharyngitis (Infections and infestations) | 26 | 25 | 15
Headache (Nervous system disorders) | 24 | 15 | 18
Nausea (Gastrointestinal disorders) | 45 | 17 | 56
Diarrhoea (Gastrointestinal disorders) | 42 | 20 | 21
Vomiting (Gastrointestinal disorders) | 15 | 7 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.